CLINICAL TRIAL: NCT00906945
Title: Chemosensitization With Plerixafor Plus G-CSF in Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Chemosensitization With Plerixafor Plus G-CSF in Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0910 / 201106039
Record Dates: First submitted 2009-05-13; First posted 2009-05-21 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: stem cell mobilization; chemosensitization; CXCR4; SDF-1; CXCL-12
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; plerixafor; Mitoxantrone; Etoposide; etoposide phosphate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Dose Level 1 (Experimental): * G-CSF 10 mcg/kg SQ on Days 1-8
  * Plerixafor 240 mcg/kg/d IV qd
  * Mitoxantrone 8 mg/m2/day IV once over 30 minutes daily on days 4-8
  * Etoposide 100 mg/m2/day IV once over 60 minutes daily on days 4-8
  * Cytarabine 1000 mg/m2/day IV once over 60 minutes daily on days 4-8
  Interventions: Drug: G-CSF; Drug: Plerixafor; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine
- Dose Level 2 (Experimental): * G-CSF 10 mcg/kg SQ on Days 1-8
  * Plerixafor 320 mcg/kg/d IV qd
  * Mitoxantrone 8 mg/m2/day IV once over 30 minutes daily on days 4-8
  * Etoposide 100 mg/m2/day IV once over 60 minutes daily on days 4-8
  * Cytarabine 1000 mg/m2/day IV once over 60 minutes daily on days 4-8
  Interventions: Drug: G-CSF; Drug: Plerixafor; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine
- Dose Level 3 (Experimental): * G-CSF 10 mcg/kg SQ on Days 1-8
  * Plerixafor 420 mcg/kg/d IV qd
  * Mitoxantrone 8 mg/m2/day IV once over 30 minutes daily on days 4-8
  * Etoposide 100 mg/m2/day IV once over 60 minutes daily on days 4-8
  * Cytarabine 1000 mg/m2/day IV once over 60 minutes daily on days 4-8
  Interventions: Drug: G-CSF; Drug: Plerixafor; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine
- Dose Level 4 (Experimental): * G-CSF 10 mcg/kg SQ on Days 1-8
  * Plerixafor 560 mcg/kg/d IV qd
  * Mitoxantrone 8 mg/m2/day IV once over 30 minutes daily on days 4-8
  * Etoposide 100 mg/m2/day IV once over 60 minutes daily on days 4-8
  * Cytarabine 1000 mg/m2/day IV once over 60 minutes daily on days 4-8
  Interventions: Drug: G-CSF; Drug: Plerixafor; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine
- Dose Level 5 (Experimental): * G-CSF 10 mcg/kg SQ on Days 1-8
  * Plerixafor 750 mcg/kg/d IV qd
  * Mitoxantrone 8 mg/m2/day IV once over 30 minutes daily on days 4-8
  * Etoposide 100 mg/m2/day IV once over 60 minutes daily on days 4-8
  * Cytarabine 1000 mg/m2/day IV once over 60 minutes daily on days 4-8
  Interventions: Drug: G-CSF; Drug: Plerixafor; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine
- MTD - Phase II (Experimental): * G-CSF MTD determined in Phase 1 SQ on Days 1-8
  * Plerixafor MTD determined in Phase 1 mcg/kg/d IV qd
  * Mitoxantrone 8 mg/m2/day IV once over 30 minutes daily on days 4-8
  * Etoposide 100 mg/m2/day IV once over 60 minutes daily on days 4-8
  * Cytarabine 1000 mg/m2/day IV once over 60 minutes daily on days 4-8
  Interventions: Drug: G-CSF; Drug: Plerixafor; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine

INTERVENTIONS:
Drug: G-CSF
  Other Names: filgrastim; Neupogen
Drug: Plerixafor
  Other Names: AMD3100; Mozobil
Drug: Mitoxantrone
  Other Names: Novantrone
Drug: Etoposide
  Other Names: VP-16; Vepesid; Etopophos
Drug: Cytarabine
  Other Names: Ara-C; Cytosar

SUMMARY:
This study is designed to test the combination of Plerixafor with G-CSF for chemosensitization in patients with relapsed or refractory AML.

DETAILED DESCRIPTION:
In this study, we are seeking to target the leukemia microenvironment to overcome disease resistance. We hypothesize that by disrupting the interaction of leukemic blasts with the bone marrow microenvironment, we may sensitize leukemic blasts to the effects of cytotoxic chemotherapy. In this study, we seek to maximize blockage of the SDF-1/CXCR4 axis through the following:

1. Addition of G-CSF, which down regulates SDF-1 expression and acts synergistically with plerixafor in stem cell mobilization
2. Intravenous instead of subcutaneous dosing of plerixafor to improve kinetics of administration.
3. Dose escalation of plerixafor and twice daily dosing to maintain maximum CXCR4 blockade.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myeloid leukemia diagnosed by WHO criteria with one of the following:

   * Primary refractory disease following no more than 2 cycles of induction chemotherapy
   * First relapse with no prior unsuccessful salvage chemotherapy
2. Age between 18 and 70 years old
3. ECOG performance status ≤ 3
4. Adequate organ function defined as:

   * Calculated creatinine clearance ≥ 50 ml/min
   * AST, ALT, total bilirubin ≤ 2 x ULN except when in the opinion of treating physician is due to direct involvement of leukemia (eg. hepatic infiltration or biliary obstruction due to leukemia)
   * Left ventricular ejection fraction of ≥ 40% by MUGA scan or echocardiogram
5. Are surgically or biologically sterile or willing to practice acceptable birth control, as follows:

   * Females of child bearing potential must agree to abstain from sexual activity or to use a medically approved contraceptive measure/regimen during and for 3 months after the treatment period. Women of child bearing potential must have a negative serum or urine pregnancy test at the time of enrollment. Acceptable methods of birth control include oral contraceptive, intrauterine device (IUD), transdermal/implanted or injected contraceptives and abstinence.
   * Males must agree to abstain from sexual activity or agree to utilize a medically approved contraception method during and for 3 months after the treatment period
6. Able to provide signed informed consent prior to registration on study

Exclusion Criteria:

1. Acute promyelocytic leukemia (AML with t(15;17)(q22;q11) and variants)
2. Peripheral blood blast count ≥ 20 x 103 /mm3
3. Active CNS involvement with leukemia
4. Previous treatment with MEC or other regimen containing both mitoxantrone and etoposide
5. Pregnant or nursing
6. Received any other investigational agent or cytotoxic chemotherapy (excluding hydroxyurea) within the preceding 2 weeks
7. Received colony stimulating factors filgrastim or sargramostim within 1 week or pegfilgrastim within 2 weeks of study
8. Severe concurrent illness that would limit compliance with study requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey L. Uy, M.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 02/04/2011 and closed to participant enrollment on 08/19/2013.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | MTD - Phase II
Started | 3 | 3 | 3 | 7 | 7 | 16
Completed | 3 | 3 | 3 | 6 | 6 | 14
Not Completed | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Found to be not eligible | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 5 (Includes MTD-Phase II): * G-CSF 10 mcg/kg SQ on Days 1-8
  * Plerixafor 750 mcg/kg/d IV qd
  * Mitoxantrone 8 mg/m2/day IV once over 30 minutes daily on days 4-8
  * Etoposide 100 mg/m2/day IV once over 60 minutes daily on days 4-8
  * Cytarabine 1000 mg/m2/day IV once over 60 minutes daily on days 4-8
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 (Includes MTD-Phase II) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 20 | 35
Age, Continuous [Median (Full Range); unit: years] | 63 [59 to 65] | 47 [43 to 50] | 64 [24 to 67] | 54 [34 to 59] | 56 [29 to 70] | 56 [24 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 4 | 8 | 17
  Male | 1 | 1 | 2 | 2 | 12 | 18
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 6 | 20 | 35

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose of Plerixafor Plus G-CSF When Combined With MEC
Time Frame: Completion of Phase I enrollment (17 months)
Population: Number of participants analyzed is the number of participants enrolled in the Phase I portion of the study.
Measure: Number; unit: mcg/kg/day
Arm/Group | Phase I (Includes Levels 1-5)
Number analyzed (Participants) | 21
mcg/kg/day | 750

2. Primary Outcome: Phase II: Complete Response Rate (CR+CRi)
Description: * Morphologic complete remission (CR): Defined as morphologic leukemia-free state, including <5% blasts in BM aspirate with marrow spicules and a count of > 200 nucleated cells and no blasts with Auer rods, no persistent extramedullary disease, ANC > 1,000/mm3, platelet count > 100,000/mm3.
  * Morphologic complete remission with incomplete blood count recovery (CRi): Defined as CR with the exception of neutropenia <1,000/mm3 or thrombocytopenia <100,000/mm3.
Time Frame: 45 days
Population: Only patients enrolled in Phase 2 portion were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Phase II (MTD)
Number analyzed (Participants) | 20
percentage of participants | 30

3. Secondary Outcome: Phase I and Phase II: Safety and Tolerability of Regimen as Measured by Grade and Frequency of Adverse Events Exceeding 10% in Total Frequency
Time Frame: 30 days following end of treatment
Measure: Number; unit: number of events
Arm/Group | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35
number of events
  Anemia | 0 | 4 | 9 | 0 | 0
  Febrile neutropenia | 0 | 0 | 20 | 0 | 0
  Abdominal pain | 6 | 0 | 1 | 0 | 0
  Constipation | 5 | 2 | 0 | 0 | 0
  Diarrhea | 7 | 6 | 0 | 0 | 0
  Gastroesophageal reflux disease | 1 | 5 | 0 | 0 | 0
  Mucositis oral | 2 | 3 | 1 | 0 | 0
  Nausea | 21 | 3 | 0 | 0 | 0
  Vomiting | 12 | 0 | 1 | 0 | 0
  Chills | 5 | 0 | 0 | 0 | 0
  Edema-limbs | 5 | 1 | 0 | 0 | 0
  Fatigue | 9 | 2 | 1 | 0 | 0
  Fever | 6 | 4 | 0 | 0 | 0
  Non-cardiac chest pain | 1 | 2 | 1 | 0 | 0
  Pain | 2 | 2 | 0 | 0 | 0
  Bacteremia | 0 | 0 | 4 | 0 | 0
  Lung infection | 0 | 1 | 5 | 0 | 2
  Sepsis | 0 | 0 | 0 | 4 | 4
  Activated partial thromboplastin time prolonged | 5 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased | 3 | 0 | 1 | 0 | 0
  Alkaline phosphatase increased | 3 | 1 | 0 | 0 | 0
  Aspartate aminotransferase increased | 4 | 0 | 0 | 0 | 0
  Blood bilirubin increased | 2 | 3 | 1 | 0 | 0
  INR increased | 7 | 0 | 0 | 0 | 0
  Neutrophil count decreased | 0 | 0 | 0 | 7 | 0
  Platelet count decreased | 0 | 0 | 0 | 15 | 0
  White blood cell count decreased | 0 | 0 | 0 | 16 | 0
  Anorexia | 4 | 2 | 0 | 0 | 0
  Hypoalbuminemia | 3 | 6 | 0 | 0 | 0
  Hypocalcemia | 2 | 11 | 0 | 0 | 0
  Hypokalemia | 5 | 2 | 2 | 2 | 0
  Hypomagnesemia | 7 | 0 | 0 | 0 | 0
  Hyponatremia | 4 | 0 | 1 | 0 | 0
  Bone pain | 4 | 2 | 2 | 0 | 0
  Dizziness | 4 | 1 | 0 | 0 | 0
  Headache | 7 | 6 | 1 | 0 | 0
  Paresthesia | 4 | 1 | 0 | 0 | 0
  Insomnia | 5 | 2 | 0 | 0 | 0
  Proteinuria | 3 | 1 | 0 | 0 | 0
  Cough | 3 | 2 | 0 | 0 | 0
  Dyspnea | 3 | 3 | 0 | 0 | 0
  Pneumonitis | 1 | 3 | 0 | 0 | 1
  Rash maculo-papular | 3 | 3 | 0 | 0 | 0
  Hypotension | 4 | 4 | 2 | 0 | 0

4. Secondary Outcome: Time to Hematologic Recovery as Measured by Time to Neutrophil Recovery
Description: -Neutrophil recovery is defined as absolute neutrophil count (ANC) >= 500/mm^3
Time Frame: Up to 62 days after treatment
Population: All participants enrolled in the study (both Phase I or Phase II) who had a CR/CRi whose ANC was >=500/mm^3 were evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 9
days | 38 [21 to 62]

5. Secondary Outcome: Time to Hematologic Recovery as Measured by Time to Neutrophil Recovery
Description: -Neutrophil recovery is defined as absolute neutrophil count >= 1000/mm^3
Time Frame: Up to 62 days after treatment
Population: All participants enrolled in the study (both Phase I or Phase II) who had a CR/CRi whose ANC was >=1000/mm^3 were evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 8
days | 40 [23 to 62]

6. Secondary Outcome: Time to Hematologic Recovery as Measured by Time to Platelet Recovery
Description: -Platelet recovery is defined as platelets >= 50,000/mm^3
Time Frame: Up to 62 days after treatment
Population: All participants enrolled in the study (both Phase I or Phase II) who had CR whose platelets were >=50,000/mm^3 were evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 9
days | 32 [27 to 62]

7. Secondary Outcome: Time to Hematologic Recovery as Measured by Time to Platelet Recovery
Description: -Platelet recovery is defined as platelets >= 100,000/mm3
Time Frame: Up to 62 days after treatment
Population: All participants enrolled in the study (both Phase I or Phase II) who had a CR whose platelets were >=100,000/mm^3 were evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 7
days | 32 [30 to 62]

8. Secondary Outcome: Characterize the Mobilization of Leukemic Cells With Plerixafor Plus G-CSF as Measured by Fold Change in White Blood Cells
Time Frame: 6 hours after plerixafor
Population: 31 patients were evaluable for this outcome measure (3 patients were never treated due to being ineligible and 1 patient never treated due to physician decision). The remaining 4 patients did not have usable peripheral blood samples for this outcome measure.
Measure: Mean (Standard Deviation); unit: fold change in white blood cells
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 31
fold change in white blood cells | 4.6 (3.6)

9. Secondary Outcome: Characterize the Mobilization of Leukemic Cells With Plerixafor Plus G-CSF as Measured by Fold Change in AML Blast Count
Time Frame: 6 hours after plerixafor
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: fold change in AML blast count
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 31
fold change in AML blast count | 9.4 (11.6)

10. Secondary Outcome: Characterize the Effects of Plerixafor Plus G-CSF on Fold Change in CXCR4 Clone 1D9 Relative Mean Fluorescent Intensity
Time Frame: 6 hours after plerixafor
Population: 29 patients were evaluable for this outcome measure (3 patients were never treated due to being ineligible and 1 patient never treated due to physician decision). The remaining 6 patients did not have usable peripheral blood samples for this outcome measure.
Measure: Mean (Standard Deviation); unit: fold change in CXCR4 clone 1D9
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 29
fold change in CXCR4 clone 1D9 | 8.0 (13.2)

11. Secondary Outcome: Characterize the Effects of Plerixafor Plus G-CSF on Fold Change in CXCR4 Clone 12G5 Relative Mean Fluorescent Intensity
Time Frame: 6 hours after plerixafor
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: fold change in CXCR4 clone 1D9
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 29
fold change in CXCR4 clone 1D9 | 0.9 (0.9)

12. Secondary Outcome: Time to Progression
Description: Recurrence / morphologic relapse: Defined as reappearance of blasts in the blood or the finding of > 5% blasts in the BM, not attributable to any other cause. New dysplastic changes are considered a relapse. If there are no blasts in the peripheral blood and 5-19% blasts in the BM, the BM biopsy and aspirate should be repeated in > 1 week to confirm relapse.
Time Frame: 2 years
Population: Data was not collected for this outcome measure. Progression is very hard to define acute myeloid leukemia and including it as a pre-specified secondary outcome measure in the protocol was an oversight.
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Time to Treatment Failure
Time Frame: 8 days
Population: Data was not collected for this outcome measure. It is not well defined in the literature as when to measure treatment failure. Relapse free survival is a better way to measure response duration (this outcome measure was added to the results).
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 0

14. Secondary Outcome: Overall Survival
Description: Overall survival: Defined as the date of first dose of study drug to the date of death from any cause.
Time Frame: Median follow-up was 34.6 months
Measure: Median (Full Range); unit: days
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 35
days | 227 [13 to 1633]

15. Post Hoc Outcome: Relapse Free-survival Rate
Time Frame: 2 years
Population: All participants enrolled in the study (both Phase I or Phase II) who had a CR/CRi were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Phase I and Phase II Participants
Number analyzed (Participants) | 9
percentage of participants | 75

ADVERSE EVENTS:
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | MTD - Phase II
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 0/3 | 2/6 | 2/6 | 2/14
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6 | 6/6 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Dose Level 4 (N=6) | Dose Level 5 (N=6) | MTD - Phase II (N=14)
Body pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac troponin increased (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 1
Subdural hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Dose Level 4 (N=6) | Dose Level 5 (N=6) | MTD - Phase II (N=14)
Abdominal cramping (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2 | 0 | 1 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 3
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 2 | 9
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Fungemia - Candida parapsilosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bacteremia - Corynebacterium Species (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bacteremia - Klebsiella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bacteremia - Staphylococcus epidermis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bacteremia - Streptococcus agalactiae (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 3
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 3 | 0
Chills (General disorders) | 1 | 0 | 1 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2 | 3 | 2 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 2 | 1
Double uterus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dysesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Edema: limbs (General disorders) | 0 | 0 | 1 | 2 | 1 | 2
Enlarged bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 2 | 1 | 4 | 2 | 1
Febrile neutropenia (Infections and infestations) | 3 | 2 | 0 | 2 | 4 | 8
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fever (General disorders) | 0 | 0 | 3 | 5 | 1 | 1
Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Graft versus host disease (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 4 | 3 | 3
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 2 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 5 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 2 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 4
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 1 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
INR increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 4
Inclusion cyst - mid thoracic back (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Increased creatinine (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2 | 1 | 3
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lip infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 3
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 5 | 5 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 1 | 0 | 4
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 1 | 1 | 0
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 2 | 1 | 0
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 2 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Perirectal abscess (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Perirectal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 2 | 1 | 1 | 0 | 2 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Pleural hemmorhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2 | 2
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Sinus pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 2
Skin infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Subconjunctival hemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Subdural hematoma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Submandibular mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 3 | 3 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 2 | 0 | 1 | 0 | 2 | 11
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes